CLINICAL TRIAL: NCT06037252
Title: A Phase 2, Randomized, Double-blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Investigational Tirzepatide Doses in Participants With Type 2 Diabetes and Obesity
Brief Title: A Study of Investigational Tirzepatide (LY3298176) Doses in Participants With Type 2 Diabetes and Obesity
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18739; I8F-MC-GPIT (Other: Eli Lilly and Company); 2023-504561-24-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases; Overnutrition; Nutrition Disorders; Body Weight; Tirzepatide; Incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Overnutrition; Nutrition Disorders; Body Weight | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tirzepatide High Dose 1 (Experimental): Participants will receive tirzepatide subcutaneously (SC).
  Interventions: Drug: Tirzepatide
- Tirzepatide High Dose 2 (Experimental): Participants will receive tirzepatide SC.
  Interventions: Drug: Tirzepatide
- Tirzepatide (Active Comparator): Participants will receive tirzepatide SC.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide; Tirzepatide High Dose 1; Tirzepatide High Dose 2
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn more about the safety and efficacy of investigational tirzepatide doses in participants with Type 2 diabetes and obesity that are already taking metformin. The study will last for about 89 weeks.

DETAILED DESCRIPTION:
The study will include a screening period of up to 5 weeks. The primary endpoint will be at Week 44 with a tirzepatide extension until week 80. A safety follow up will be performed approximately 4 weeks after end of treatment.

ELIGIBILITY:
Inclusion Criteria

* Have a Body Mass Index (BMI) ≥35 kilogram/square meter (kg/m²) at screening.
* Have had stable body weight (±5%) during the 90 days preceding screening.
* Have been diagnosed with Type 2 Diabetes (T2D).
* Have been on a stable treatment of metformin only at least 90 days preceding screening and between screening and randomization with the minimum effective dose of ≥1500 milligram (mg)/day.

Exclusion Criteria:

* Have Type 1 Diabetes (T1D), history of ketoacidosis or hyperosmolar state/coma, or any other types of diabetes except T2D.
* Have had 1 or more episode of severe hypoglycemia and/or 1 or more episode of hypoglycemia unawareness within 6 months prior to screening.
* Are currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema.
* Have a prior or planned surgical treatment for obesity.
* Use products intended for weight loss including prescription drugs, over the counter (OTC) drugs, and herbal preparations, within 3 months prior to screening.
* Have renal impairment measured as estimated glomerular filtration rate (eGFR) <45 milliliter/min (mL/min)/1.73 m².
* Have any of the following cardiovascular (CV) conditions within 2 months prior to screening.

  * acute myocardial infarction.
  * cerebrovascular accident (stroke).
  * unstable angina .
  * hospitalization due to congestive heart failure, or
  * coronary artery revascularization.
* Have a family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia (MEN) syndrome Type 2.
* Have a history of chronic or acute pancreatitis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Body Weight | Baseline (Week 0), Week 44

SECONDARY OUTCOMES:
Change from Baseline in HbA1c | Baseline (Week 0), Week 44
Change from Baseline in HbA1c | Baseline (Week 24), Week 80
Percent Change from Baseline in Body Weight | Baseline (Week 24), Week 80
Absolute Change from Baseline in Body Weight | Baseline (Week 0), Week 44
Absolute Change from Baseline in Body Weight | Baseline (Week 24), Week 80
Change from Baseline in Body Mass Index (BMI) | Baseline (Week 0), Week 44
Change from Baseline in BMI | Baseline (Week 24), Week 80
Change from Baseline in Waist Circumference | Baseline (Week 0), Week 44
Change from Baseline in Waist Circumference | Baseline (Week 24), Week 80
Percentage of Participants Achieving ≥15% Body Weight Reduction | Baseline (Week 0), Week 44
Percentage of Participants Achieving ≥15% Body Weight Reduction | Baseline (Week 0), Week 80
Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC) | Baseline through Week 44
  Steady State Area Under the Concentration Time Curve (AUC) presented as a single average measure of AUC across the time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- United States (20):
  - Medical Advancement Centers of Arizona, Phoenix, Arizona
  - John Muir Physician Network Research Center, Concord, California
  - Care Access - Sacramento, Sacramento, California
  - Care Access - Aurora, Aurora, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Retreat Medical Research, Miami, Florida
  - American Research Centers of Florida, Pembroke Pines, Florida
  - Alta Pharmaceutical Research Center, Norcross, Georgia
  - AGILE Clinical Research Trials, LLC, Sandy Springs, Georgia
  - Northwestern University, Chicago, Illinois
  - Qualmedica Research, LLC, Evansville, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Accellacare - Wilmington - 1917 Tradd Court, Wilmington, North Carolina
  - Velocity Clinical Research, Mt. Auburn, Cincinnati, Ohio
  - Summit Headlands, Portland, Oregon
  - Clinical Research Associates Inc, Nashville, Tennessee
  - Juno Research, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
- Argentina (5):
  - CEDIC, CABA, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro Médico Viamonte, Buenos Aires, Buenos Aires F.D.
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires, Buenos Aires F.D.
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
- Mexico (6):
  - Centro de Investigacion Cardiovascular y Metabólica, Tijuana, Estado de Baja California
  - Virgen Cardiovascular Research SC, Guadalajara, Jalisco
  - Cryptex Investigación Clínica S.A. de C.V., Cuauhtémoc, Ciudad de México, Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero, Tamaulipas
- Turkey (Türkiye) (9):
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Kadıköy, Istanbul
  - Baskent Universitesi Adana Dr. Turgut Noyan Uygulama ve Arastirma Merkezi, Adana
  - Akdeniz Universitesi Hastanesi, Antalya
  - Uludag Universitesi, Bursa
  - Dicle Üniversitesi, Diyarbakır
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - Acibadem Universitesi Atakent Hastanesi, Istanbul
  - Marmara Universitesi Pendik Egitim Arastirma Hastanesi, Istanbul
  - Ondokuz Mayıs Universitesi, Samsun

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: ata are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Investigational Tirzepatide (LY3298176) Doses in Participants With Type 2 Diabetes and Obesity — https://trials.lilly.com/en-US/trial/422915